CLINICAL TRIAL: NCT02312362
Title: HFDS ab Interno - to Compare Intraocular Pressure (IOP) Lowering Effect of Combined High Frequency Deep Sclerotomy ab Interno (HFDS ab Interno) With Phacoemulsification and Phacoemulsification Alone, in Primary Open Angle Glaucoma Patients
Brief Title: High Frequency Deep Sclerotomy (HFDS) ab Interno a Combination Surgical Intervention Using Cataract Surgery to Lower IOP
Acronym: HFDS_abinterno
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oertli Instrumente AG (Industry)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFDS_PS_v9
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Cataract; Glaucoma; POAG
Keywords: HFDS; ab interno; MIGS; surgery
MeSH Terms: conditions — Cataract; Glaucoma | interventions — rhoA GTP-Binding Protein; Phacoemulsification; Cataract Extraction

ARMS (2):
- Combined sclerotomy ab interno and phaco (Experimental): Combined sclerotomy ab interno and phacoemulsification with IOL implantation
  Interventions: Procedure: Combined sclerotomy ab interno and phaco
- Phacoemulsification with IOL implantation (Active Comparator): Phacoemulsification with IOL implantation
  Interventions: Procedure: Phacoemulsification with IOL implantation

INTERVENTIONS:
Procedure: Combined sclerotomy ab interno and phaco
  Other Names: High Frequency Deep Sclerotomy (=HFDS); HFDS; STT (formerly); abee tip; Cataract surgery combined with HFDS
  Arms: Combined sclerotomy ab interno and phaco
Procedure: Phacoemulsification with IOL implantation
  Other Names: Phacoemulsification; Phaco; Cataract Surgery
  Arms: Phacoemulsification with IOL implantation

SUMMARY:
Objective:

To compare intraocular pressure lowering effect of combined sclerotomy ab interno with phacoemulsification and phacoemulsification alone, in primary or secondary open angle glaucoma patients.

Study design:

Prospective, randomized, case- control interventional surgical trial

ELIGIBILITY:
Inclusion Criteria:

Patients suffering from primary open-angle glaucoma (POAG) inadequately controlled with maximum tolerated medical therapy and who will be treated with cataract surgery.

Exclusion Criteria:

* One eyed patients
* Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits
* The presence of extreme narrow angle with complete or partial closure in either eye, except for occludable angles treated with a patent iridectomy
* Any abnormality preventing reliable applanation tonometry, any opacity or patient uncooperativeness that would restrict adequate examination of the ocular fundus or anterior chamber of either eye
* The risk of visual field or visual acuity worsening as a consequence of participation in the trial, in the investigator's opinion
* Any clinically significant, serious, or severe medical or psychiatric condition; any condition that, in the investigator's opinion, would interfere with optimal participation in the study or present a special risk to the patient
* Participation in any other investigational study within 30 days prior to baseline visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Baseline screening till 3 year post-op
visual acuity | Baseline screening till 3 year post-op
decrease in anti glaucoma medications | Baseline screening till 3 year post-op

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Hafezi, MD, PhD, Principal Investigator — University of Geneva, Switzerland
Locations (5):
- Aswān, Egypt
- Kiel, Germany
- Mumbai, India
- Switzerland (2):
  - Geneva
  - Reinach

REFERENCES:
- [Background] Pajic B, Pajic-Eggspuehler B, Haefliger I. New minimally invasive, deep sclerotomy ab interno surgical procedure for glaucoma, six years of follow-up. J Glaucoma. 2011 Feb;20(2):109-14. doi: 10.1097/IJG.0b013e3181dddf31. PMID 20520572